CLINICAL TRIAL: NCT07281157
Title: The Combination of Irinotecan Liposome, Capecitabine and Enlansubemab Embedded in Short-course Radiotherapy as Neoadjuvant Therapy for Locally Advanced Rectal Cancer: a Prospective, Single-center and Single-arm Study
Brief Title: Irinotecan Liposome Plus Capecitabine and Enronsubemab Combined With Short-course Radiotherapy for Neoadjuvant Treatment of Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DNY-CRC-TJ04
Record Dates: First submitted 2025-12-01; First posted 2025-12-15 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-10

CONDITIONS: Advanced Colorectal Cancer
MeSH Terms: interventions — irinotecan sucrosofate; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan Liposome, Capecitabine, and Enlansubemab Plus Short-Course Radiotherapy (Experimental)
  Interventions: Drug: Irinotecan Liposome, Capecitabine, and Enlansubemab Plus Short-Course Radiotherapy

INTERVENTIONS:
Drug: Irinotecan Liposome, Capecitabine, and Enlansubemab Plus Short-Course Radiotherapy — Phase One: Induction immunotherapy Irinotecan liposome: 50mg/m2, ivgtt, d1; Capecitabine: 825mg/m2, po, bid, d1-10; Enlangsumab: 240mg, ivgtt, d1. Repeat every two weeks for two treatment cycles
  Phase Two: Short-course radiotherapy Short-course radiotherapy: 5x5Gy, once a day, 5Gy each time, for 5 consecutive days. After radiotherapy, rest for 7 to 14 days before starting consolidation immunotherapy. After radiotherapy, conduct imaging evaluations of tumor remission.
  Phase Three: Consolidation of chemotherapy-free treatment Irinotecan liposome: 50mg/m2, ivgtt, d1; Capecitabine: 825mg/m2, po, bid, d1-10; Enlangsumab: 240mg, ivgtt, d1. Repeat every two weeks for four treatment cycles
  Phase Four: W&W

SUMMARY:
This is a prospective, single-center, single-arm study on the combination regimen of irinotecan liposome, capecitabine and enronsubemab embedded in short-course radiotherapy as neoadjuvant therapy for locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-75 years old;
2. rectal adenocarcinoma confirmed by histology and/or cytology;
3. locally advanced rectal cancer cT3-4 or N+ confirmed by baseline examination (AJCC/UICC TNM staging (8th edition, 2017);
4. Distance from lower margin to anal margin ≤ 10 cm;
5. Patients with at least one assessable lesion according to RECIST1.1 criteria;
6. ECOG 0-1;
7. the expected survival time was more than 12 months;
8. had not received anti-tumor treatment for rectal cancer after diagnosis, including radiotherapy, chemotherapy, surgery, etc.
9. Bone marrow function: absolute neutrophil count (ANC) ≥1.5×109/L, hemoglobin ≥90g/dL, platelet (PLT) ≥100×109/L, white blood cell (WBC) ≥3.0×109/L;
10. Liver function: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) ≤2.5 times the upper limit of normal (ULN), if there is liver metastasis ≤5×ULN, total bilirubin <1.5 ULN;
11. Renal function: serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (CCr) ≥60mL/min (according to Cockcroft-Gault formula);
12. Coagulation function: prothrombin time (PT), activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤1.5×ULN;
13. exclude active or suspected infection;
14. non-pregnant or lactating women; Women/men of childbearing age should use effective contraception during the study and for 6 months after the end of study treatment;
15. The patients had good compliance, understood the research process of this study, and signed the written informed consent.

Exclusion Criteria:

1. patients with other malignant tumors (except cured carcinoma in situ and basal cell carcinoma) in the past 5 years;
2. patients with mismatch repair deficiency (dMMR) or microsatellite instability high (MSI-H);
3. obvious clinical bleeding symptoms or obvious bleeding tendency within 3 months before treatment (bleeding > 30 mL within 3 months, hematemesis, melena, hematochezia), hemoptysis (fresh blood > 5 mL within 4 weeks), etc. Or treatment for a venous/venous thrombotic event within the previous 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism; Long-term anticoagulation with warfarin or heparin or long-term antiplatelet therapy (aspirin ≥300 mg/ day or clopidogrel ≥75 mg/ day) may be required.
4. extensive distant metastasis (e.g., peritoneal metastasis, multiple bone/brain metastases);
5. patients who had used potent CYP3A4 inducers at the same time within 3 weeks before the first dose, or had used potent CYP3A4 inhibitors or potent UGT1A1 inhibitors within 3 weeks before the first dose;
6. patients who underwent major organ surgery (excluding needle biopsy, central venous catheterization, port catheterization, stent placement to relieve biliary obstruction, percutaneous hepatobiliary drainage, cholecystostomy) or elective surgery within 4 weeks before treatment;
7. tumor invasion of large vascular structures, such as pulmonary artery, superior vena cava or inferior vena cava, and there is a high risk of bleeding according to the investigator's judgment;
8. Active heart disease (including myocardial infarction, severe/unstable angina) within 6 months before treatment. Echocardiography showed that the left ventricular ejection fraction was less than 50% and the arrhythmia was not well controlled.
9. have hypertension that is not well controlled with antihypertensive medication (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg);
10. subjects with active infection or fever of unknown origin >38.5 degrees during screening or before the first dose of medication (according to the investigator's assessment, subjects with fever due to cancer could be enrolled);
11. subjects with congenital or acquired immunodeficiency, such as HIV infection or active hepatitis (transaminase did not meet the inclusion criteria, hepatitis B reference: HBV DNA≥1000 IU/ml; hepatitis C reference: HCV RNA≥1000 IU/ml); Chronic hepatitis B virus carriers, HBV DNA < 2000 IU/ml, must receive antiviral therapy at the same time during the trial.
12. any other medical condition, clinically significant metabolic abnormality, physical examination abnormality, or laboratory abnormality where there is reason to suspect that the patient has a disease or condition (such as having seizures requiring treatment) that would be inappropriate for the study drug, in the investigator's judgment, or that would affect interpretation of the study results or place the patient at high risk;
13. intestinal obstruction (except incomplete intestinal obstruction requiring only enteral nutrition); Subjects at risk of intestinal perforation (including, but not limited to, a history of acute diverticulitis, abdominal abscess, or abdominal cancer); 14 History of wide bowel resection (partial colectomy or wide small bowel resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.

(15) received any other antibodies/drugs (including PD-1, PD-L1, PD-L2, CTLA-4, OX40, C137 inhibitors, etc.) acting on T cell costimulation or checkpoint pathway.

(16) patients with CTCAE 5.0 grade ≥ 3 immune-related adverse events (AE) after immunotherapy.

(17) patients receiving glucocorticoid (prednisone >10mg/ day or equivalent dose of other drugs of the same kind) or other immunosuppressive therapy for some condition within 14 days before the first dose of the drug.

(18) participated in other clinical investigators within 4 weeks before enrollment; (19) a documented history of allergy to study drugs, including enlansubemab, capecitabine, liposome-irinotecan, and any component of the drug; (20) pregnant or lactating female subjects; Patients deemed by the investigator to be ineligible for trial participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2032-04-30 (Estimated)

PRIMARY OUTCOMES:
Complete response plus pathological complete response | 1 year
  Through imaging examinations such as CT, MRI or PET-CT, it was confirmed that all visible tumor lesions had completely disappeared and remained there for at least 4 weeks. After surgical resection of the tumor tissue, no residual cancer cells (including the primary lesion and lymph nodes) were found under microscopic examination.

SECONDARY OUTCOMES:
Progression-free survival | 2 year
  The time from randomization to disease progression or death
OS | 3 year
  The period from the time a patient randomly receives treatment until death due to any cause.
Adverse Event | 3 year
  All adverse medical events that occurred after the subjects accepted the trial protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China